CLINICAL TRIAL: NCT06131346
Title: Identification, Clinical Characterization, and Prognosis of Anti-IgLON5 Disease
Brief Title: Clinical Characterization and Outcome of Anti-IgLON5 Disease
Acronym: ICP-IGLON5
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1173
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Anti-IgLON5 Disease
Keywords: Anti-IgLON5 disease, autoimmune encephalitis, neural antibodies
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with anti-IgLON5 antibodies: Adults patients who tested positive for anti-IgLON5 antibodies in the French Reference centre of Autoimmune Encephalitis
  Interventions: Other: Evaluation of clinical and paraclinical data.

INTERVENTIONS:
Other: Evaluation of clinical and paraclinical data. — Retrospective data collection from available medical files of patient.

SUMMARY:
Anti-IgLON5 disease is a neurological disorder associated with antibodies to IgLON5, a neuronal cell adhesion protein of unknown function. Most patients develop a combination of significant sleep disturbances (non-rapid eye movement (NREM) and rapid eye movement parasomnias with obstructive sleep apnoea), bulbar dysfunction (dysarthria, dysphagia, vocal cord paralysis or episodes of respiratory failure) and gait instability. Early autopsy studies showed deposits of phosphorylated tau protein mainly in neurons of the brainstem tegmentum, suggesting a primary neurodegenerative disease. However, the results of subsequent studies have provided increasing support for an immune-mediated pathogenesis. First, there is a strong association with the human leukocyte antigen (HLA) haplotype DRB1*10:01-DQB1*05 : 01, which is present in ~60% of patients (compared to 2% in the normal population); secondly, recent autopsy studies have shown the absence of abnormal tau deposits; and thirdly, in live neurons in culture, IgLON5 antibodies cause irreversible loss of surface IgLON5 clusters and cytoskeletal changes such as dystrophic neurites and axonal bulges. Together, these studies suggest that antibody-mediated disruption of IgLON5 function leads to neurofilament and cytoskeletal alterations that can potentially result in tau accumulation.

Over the last two years, an increase in diagnoses of anti-IgLON5 disease has been observed in the French Reference centre of Autoimmune Encephalitis. This could be related to a better knowledge of the disease, or to other yet unknown factors. Clinical characterisation of these patients is essential to understand the underlying reasons for the increase in diagnoses and to improve knowledge of this disease. Furthermore, the response of these patients to immunosuppressive drugs and the long-term prognosis remain unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 ans
* Anti-IgLON5 antibody positivity

Exclusion Criteria:

- Lack of clinical data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients tested positive for anti-IgLON5 antibodies.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of IGLON5 disorder | At baseline
  Prevalence of :
  * Sleeping disorders
  * Respiratory dosorders
  * Cognitive disorders
  * Abnormal movements

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France